CLINICAL TRIAL: NCT01930032
Title: Pathogenic Mechanisms in Clostridium Difficile Infection and Colitis
Brief Title: Pathogenic Mechanisms in C Diff Infection and Colitis
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Ciaran Kelly, Professor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2013P000174
Record Dates: First submitted 2013-08-20; First posted 2013-08-28 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Colonic biopsy samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All subjects

SUMMARY:
The purpose of this study is to learn more about infection by Clostridium difficile (also known as C. difficile). C. difficile is a common bacterium (a germ that may cause disease) that can live in the human gut. Some people have it without having any symptoms. In other people it can cause illness ranging from mild diarrhea to severe colitis (infection of the colon).

C. difficile makes toxins that damage the cells that line the colon. The study doctors want to find out how these toxins cause damage to the cells in the colon.

DETAILED DESCRIPTION:
The purpose of this study is to examine pathogenic mechanisms of Clostridium difficile toxin-mediated intestinal injury and inflammation. Two primary mechanisms will be examined.

* To examine the hypothesis is that microRNA expression profiles are dysregulated by Clostridium difficile toxin exposure and that dysregulation of miRNA expression plays a role in the pathogenesis of C. difficile associated diseases.
* To examine the hypothesis is that the TLR9 receptor mediates key inflammatory events in response to Clostridium difficile toxin exposure.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 yrs and less than 75 years
* Undergoing a clinically indicated colonoscopy

Exclusion Criteria:

* Known, active or recurrent colonic disease including: Clostridium difficile infection, inflammatory bowel disease, microscopic colitis, colon resection for any reason, ischemic colitis, recurrent diverticulitis, colon cancer. Note: Diverticulosis without recurrent diverticulitis, colonic adenomatous or hyperplastic polyps or colonic arteriovenous malformations will not constitute an exclusion
* Diarrhea (an average of more than 3 bowel movements per day at baseline)
* Constipation (an average of fewer than 2 bowel movements per week at baseline).
* Use of systemic steroid or systemic immunosuppressive medication
* Severe renal impairment
* Relative contraindication to colon biopsy including a bleeding diathesis or anti-coagulant use. Note: nonsteroidal antiinflammatory drug or asprin use will not constitute a contra-indication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from patients undergoing a routine screening colonoscopy at Beth Israel Deaconess Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Binding of Toxin A (and B) to TLR9 on the human colorectal epithelial cell surface | 24 hours
  As assessed by confocal fluorescence microscopy

SECONDARY OUTCOMES:
effects of a TLR9 antagonist (ODN-TTAGGG) on toxin binding | 0 hours
  The change of mean toxin fluorescence on colonocytes will be measured by confocal microscopy using quantitative image analysis software.
Binding of Toxin A (and B) to TLR9 on the human colorectal epithelial cell surface | 0 hours
  as assessed by confocal fluorescence microscopy
Binding of Toxin A (and B) to TLR9 on the human colorectal epithelial cell surface | 6 hours
  As assessed by confocal fluorescence microscopy
Effects of a TLR9 antagonist (ODN-TTAGGG) on toxin binding | 6 hours
  The change of mean toxin fluorescence on colonocytes will be measured by confocal microscopy using quantitative image analysis software.
Effects of a TLR9 antagonist (ODN-TTAGGG) on toxin binding | 24 hours
  The change of mean toxin fluorescence on colonocytes will be measured by confocal microscopy using quantitative image analysis software.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States